CLINICAL TRIAL: NCT05470582
Title: Randomized, Double-blind, Comparative, Controlled Trial of Tolerability, Safety and Immunogenicity of the Flu-M Vaccine in Children Between 6 Months and 9 Years Old
Brief Title: Trial of Tolerability, Safety and Immunogenicity of the Flu-M Vaccine in Children Between 6 Months and 9 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FLM-04-2020
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Influenza, Human; Vaccination; Infection; Vaccines
Keywords: Influenza; Flu; Vaccine; FLU-M; SPbSRIVS; Vaxigrip; Children
MeSH Terms: conditions — Influenza, Human; Infections | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flu-M, children aged 3-9 years (Experimental)
  Interventions: Biological: Flu-M, Inactivated split influenza vaccine 0.5 mL
- Vaxigrip, children aged 3-9 years (Active Comparator)
  Interventions: Biological: Vaxigrip, Inactivated split influenza vaccine 0.5 mL
- Flu-M, children aged 6-35 months (Experimental)
  Interventions: Biological: Flu-M, Inactivated split influenza vaccine 0.25 mL
- Vaxigrip, children aged 6-35 months (Active Comparator)
  Interventions: Biological: Vaxigrip, Inactivated split influenza vaccine 0.25 mL

INTERVENTIONS:
Biological: Flu-M, Inactivated split influenza vaccine 0.5 mL — Solution for intramuscular injection Сhildren were vaccinated with the Flu-M vaccine once/twice (all children were vaccinated twice with an interval of 28 days between the first vaccination and revaccination; if the child is vaccinated for the first time) intramuscularly in a dose of 0.5 mL
  Arms: Flu-M, children aged 3-9 years
Biological: Vaxigrip, Inactivated split influenza vaccine 0.5 mL — Suspension for intramuscular and subcutaneous injection Children were vaccinated with the Vaxigrip® vaccine once/twice (all children were vaccinated twice with an interval of 28 days between the first vaccination and revaccination; if the child is vaccinated for the first time) intramuscularly in a dose of 0.5 mL
  Arms: Vaxigrip, children aged 3-9 years
Biological: Flu-M, Inactivated split influenza vaccine 0.25 mL — Solution for intramuscular injection Children were vaccinated with the Flu-M vaccine twice (all children were vaccinated twice with an interval of 28 days between the first vaccination and revaccination) intramuscularly in a dose of 0.25 mL
  Arms: Flu-M, children aged 6-35 months
Biological: Vaxigrip, Inactivated split influenza vaccine 0.25 mL — Suspension for intramuscular and subcutaneous injection Children were vaccinated with the Vaxigrip® vaccine twice (all children were vaccinated twice with an interval of 28 days between the first vaccination and revaccination) intramuscularly in a dose of 0.25 mL
  Arms: Vaxigrip, children aged 6-35 months

SUMMARY:
Comparative trial of tolerability, reactogenicity, safety and immunogenicity of the Flu-M vaccine as compared to the Vaxigrip® vaccine in terms of prevention of influenza in children aged 6 months to 9 years (at the time of the first vaccination).

DETAILED DESCRIPTION:
The trial includes 2 stages (stage I, II). At stage I children aged 3-9 years will be included. Based on findings from tolerability and safety assessment in respect of the Flu-M vaccine vs. the Vaxigrip® vaccine for the first 7 days after vaccination of volunteers during Stage I, an intermediate report will be prepared. The report will be submitted to the supervisory executive authorities alongside the notice of commencement of Stage II of the trial - the continuation of trial on children aged 3-9 years and the commencement of trial on children aged between 6 months and 35 months. During Stage II, the trial for Stage I volunteers will continue in full and also children aged between 6 and 35 months will be included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* For volunteers aged 3 to 9 years:

  * Healthy children of both sexes aged 3 to 9 years (3 years 0 months 0 days - 8 years 11 months 30 days);
  * The written and dated informed consent of one of the parents for participation in the trial;
* For volunteers aged 6 to 35 months:

  * Healthy children of both genders aged 6 to 35 months, inclusive (6 months 0 days - 35 months 30 days);
  * The written and dated informed consent of one of the parents for participation in the trial;
  * The trial subject of the was born full-term, with the Apgar score of 7-10 points.
* For all volunteers:

Ability of a volunteer's parents to fulfill the requirements of the Protocol (i.e. to fill out the Patient Diary, come to visit with the volunteer).

Exclusion Criteria:

1. History of influenza (including in mothers for children aged 6 to 35 months) or previous influenza vaccination during 6 months before the trial;
2. Positive result of the SARS-CoV-2 test;
3. Vaccination of the pregnant woman in the 2nd-3rd trimester (for the age group of 6 - 35 months) with an influenza vaccine;
4. Vaccination with any vaccine less than 30 days before participating in the trial or scheduled vaccination with any vaccine within 30 days after vaccination with the trial vaccines;
5. A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter at the injection site) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination), encephalopathy;
6. Allergic reactions to vaccine components or any previous vaccination;
7. History of allergic reaction to chicken protein;
8. History of cancer, leukemia, tuberculosis, autoimmune diseases;
9. Carriage of HIV, syphilis, hepatitis B and C in the medical history, including by parents;
10. Children who received immunoglobulin products or transfusions of whole blood or its components less than 3 months before the start of the trial;
11. Long-term use (more than 14 days) of any immunomodulating medicines less than 3 months before the start of the trial;
12. Any confirmed or suspected immunosuppressive or immunodeficiency condition;
13. History of chronic diseases of the cardiovascular, bronchopulmonary, endocrine systems, blood in the acute stage (recovery less than 4 weeks before vaccination) or in the decompensation stage;
14. Children with hemophilia who may develop bleeding after intramuscular injection;
15. History of progressive neurological pathology, convulsive syndrome, afebrile convulsions;
16. History of acute infectious diseases (fever ≥ 37.5°С): recovery less than 2 weeks before vaccination;
17. Participation in another clinical trial less than 3 months before the start of the trial;
18. History of mental illness of the child and the volunteer's parents;
19. The history of the volunteer's parent being registered with a tuberculosis dispensary and/or a narcological dispensary;
20. Maternal history of drug use or alcohol abuse during pregnancy and/or breastfeeding;
21. Pronounced congenital malformations in a child;
22. Suspected developmental delay in a child.

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1066 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline seroconversion level | Days 0 (screening), 28, 56, 180 after vaccination/revaccination
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay) The upper limit of bilateral 95 % CI for the difference between seroconversion levels (seroconversion level reference vaccine - the seroconversion level trial vaccine) should not exceed 10%.
  Seroconversion ≥ 40%

SECONDARY OUTCOMES:
Change from Baseline Geometric mean titer (GMT) of antibodies | Days 0 (screening), 28 after vaccination/revaccination
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay) The upper limit of bilateral 95% CI for the GMT ratio (GMTreference vaccine/GMTtrial vaccine) should not exceed 1.5
Change from Baseline Seroconversion factor | Days 0 (screening), 28, 56, 180 after vaccination/revaccination
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay) Seroconversion factor ≥ 2.5
Change from Baseline Seroprotection rate | Days 0 (screening), 28, 56, 180 after vaccination/revaccination
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay) Seroprotection ≥ 70%
Change from Baseline Seroconversion rate for each virus strain | Days 0 (screening), 28, 56, 180 after vaccination/revaccination
  Specific anti-influenza antibodies were determined using haemagglutination inhibition assay (HI assay)
Incidence of immediate adverse events (allergic reactions) | 2 hours after vaccination/revaccination
  Anaphylaxis, Quincke's edema, Urticaria.
Incidence of local adverse events | Day 1 (2 and 5-8 hours after vaccination/revaccination), days 2-180
  Pain at the injection site at palpation, Hyperemia at the injection site, infiltrate at the injection site, Edema at the injection site, Pruritus at the injection site, Enlarged regional lymph nodes.
Incidence of systemic adverse events | Day 1 (2 and 5-8 hours after vaccination/revaccination), days 2-180
  Headache, Cough, Sore throat, Nausea, Increased sweating, Arthralgia, Myalgia, Fever, Chills, Asthenia
Incidence of severe adverse events during the trial | Day 1 (2 and 5-8 hours after vaccination/revaccination), days 2-180
Number of participants with abnormal changes in physical examination data | Days 0 (screening), 3, 7, 28, 56
  Physical examination of volunteers includes an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion; examination of skin, mucosa, eyes, oral cavity and pharynx, lungs/chest, heart/cardiovascular system, abdominal organs, nervous system, lymph nodes, musculoskeletal system.
Number of participants with abnormal changes of neurological status | Days 0 (screening), 3, 7, 28, 56
Number of participants with abnormal changes in vital signs - Blood pressure (BP) | Days 0 (screening), 3, 7, 28, 56
  BP measurements include the systolic and diastolic blood pressure.
Number of participants with abnormal changes in vital signs - Heart rate (HR) | Days 0 (screening), 3, 7, 28, 56
  HR is measured using a phonendoscope at the apex of the heart during 1 minute.
Number of participants with abnormal changes in vital signs - Respiratory rate (RR) | Days 0 (screening), 3, 7, 28, 56
  RR is counted with a hand placed on the child's chest or abdomen or by holding a stethoscope at the child's nose. The measurement is carried out during one minute.
Number of participants with abnormal changes in vital signs - Body temperature | Day 0 (screening); 10 min before, 20 min and 2 hours after vaccination; days 3, 7, 28, 56
  Measurement with a digital thermometer.
Number of participants with clinically significant abnormalities - Complete blood count (CBC) | Days 0 (screening), 3
  Hemoglobin, hematocrit, erythrocytes, leukocytes, leukocytic formula, platelets, erythrocyte sedimentation rate (ESR).
Number of participants with clinically significant abnormalities - Biochemical blood test (BBT) | Days 0 (screening), 3
  ALT, AST, LDH, alkaline phosphatase, total bilirubin, urea, glucose.
Number of participants with clinically significant abnormalities - Urinalysis | Days 0 (screening), 3
  pH, specific density, protein, glucose, erythrocytes, leukocytes.
Number of participants with abnormal changes of total IgE | Days 0 (screening), 3, 56

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, PhD, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (2):
- Russia (2):
  - LLC "Energiya zdorov'ya", Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health Care "Children's City Polyclinic No. 45" of the Nevsky District, Saint Petersburg